CLINICAL TRIAL: NCT01918280
Title: Fertility Preservation in Cases of Spermatogenesis Failure : Prospective Study for Klinefelter Syndrome With Non-mosaic Karyotype (47, XXY, Homogeneous)
Brief Title: Fertility Preservation in Cases of Klinefelter Syndrome.
Acronym: FERTIPRESERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009.576
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter Syndrome; Azoospermia; Seminal analyses; Testicular biopsy
MeSH Terms: conditions — Klinefelter Syndrome; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young group (Experimental): Patient aged 15-22 years for seminal analyses and testicular biopsy
  Interventions: Procedure: Seminal analyses and testicular biopsy
- Adult group (Other): Patient aged 23-55 years for seminal analyses and testicular biopsy
  Interventions: Procedure: Seminal analyses and testicular biopsy

INTERVENTIONS:
Procedure: Seminal analyses and testicular biopsy — Two seminal analyses spaced out 3 months followed by a testicular biopsy if the azoospermia is confirmed on semen analyses.

SUMMARY:
Klinefelter Syndrome (KS) is the most common sex chromosomal abnormalities (1/600 newborn males), and is characterized by a hypergonadism hypogonadism. Until few years ago, mostly non-mosaic KS was considered as a model of a complete male infertility although few KS (4-8%) have an oligospermia. Recent studies in adult with non-mosaic KS reported the possibility of sperm retrieval by testicular biopsy (TESE) in around 50% cases and more than some pregnancies have been obtained after TESE with Intracytoplasmic Sperm Injection (ICSI). Since 1997, more than one hundred births are described.

As some studies shown a decrease of successful sperm retrieval with the increasing of age, we plan to compare the potential of sperm retrieval between two groups "adult" (23-55 years) and "young" after the onset of puberty (15-22 years). The study will be performed by searching spermatozoa on two seminal analyses spaced out 3 months followed by a testicular biopsy if the azoospermia is confirmed on semen analyses.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter Syndrome with 47,XXY non-mosaic
* Androgenotherapy stopped since more than 6 months

Exclusion Criteria:

* Antecedent of Radiotherapy or chemotherapy
* Psychological trouble
* Treatment interfering with spermatogenesis
* Androgenotherapy non stopped

Ages: 15 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
TEsticular Sperm Extraction (TESE) | 15 months
  Improvement of sperm retrieval rate by Testicular Sperm extraction (TESE) in the "Young" group compare to "Adult" group.

SECONDARY OUTCOMES:
Androgenotherapy | 15 months
  Influence of antecedent of androgenotherapy before Testicular Sperm extraction (TESE) : treatment or not, duration of treatment
Prognosis factors | 15 months
  Identification of prognosis factors of sperm retrieval (by TESE) in the two groups "Young" and "Adult"
Histopathologist analyses | 15 months
  Histopathologist analyses of testicular biopsy in the two groups "Young" and "Adult". In the 2 groups, comparison of cases with and without sperm.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid PLOTTON, MD, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Service de Biologie de la Reproduction - CECOS - Groupe Hospitalier Pellegrin, Bordeaux
  - Service d'Endocrinologie Moléculaire et Maladies Rares, Centre de Biologie Est, Hospices Civils de Lyon, Bron
  - Service de Biologie de la Reproduction - Hôpital de la Conception, Marseille
  - Groupe de Médecine de la Reproduction - CECOS Midi-Pyrénées - Hôpital Paule de Viguier), Toulouse

REFERENCES:
- [Result] Plotton I, Giscard d'Estaing S, Cuzin B, Brosse A, Benchaib M, Lornage J, Ecochard R, Dijoud F, Lejeune H; FERTIPRESERVE group. Preliminary results of a prospective study of testicular sperm extraction in young versus adult patients with nonmosaic 47,XXY Klinefelter syndrome. J Clin Endocrinol Metab. 2015 Mar;100(3):961-7. doi: 10.1210/jc.2014-3083. Epub 2014 Nov 25. PMID 25423570
- [Result] Renault L, Labrune E, Giscard d'Estaing S, Cuzin B, Lapoirie M, Benchaib M, Lornage J, Soignon G, de Souza A, Dijoud F, Fraison E, Pral-Chatillon L, Bordes A, Sanlaville D, Schluth-Bolard C, Salle B, Ecochard R, Lejeune H, Plotton I. Delaying testicular sperm extraction in 47,XXY Klinefelter patients does not impair the sperm retrieval rate, and AMH levels are higher when TESE is positive. Hum Reprod. 2022 Oct 31;37(11):2518-2531. doi: 10.1093/humrep/deac203. PMID 36112034